CLINICAL TRIAL: NCT01527708
Title: Repeatability, Reliability and Reproducibility of Pentacam-derived Curvature and Wavefront Aberrations of Posterior Corneal Surface, in Keratoconic and Cross-linked Corneas
Brief Title: Accuracy of Curvature and Wavefront Aberrations of Posterior Corneal Surface, in Keratoconic and Post-CXL Corneas
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Lecturer, Democritus University of Thrace
Other Study IDs: 27/27-09-11
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-01

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Keratoconus Group (KCG): Keratoconus group (KCG) included patients with progressive keratoconus.
- Collagen-Cross-linking group (CXLG): Collagen-Cross-linking group (CXLG) included keratoconus patients that had been treated with uneventful corneal collagen cross-linking (CXL) at least on year prior to their enrolment in the study.
  Interventions: Procedure: Corneal Collagen Cross-linking (CXL)
- Normal Group (NG): Normal group (NG) was formed by refractive surgery candidates who visited EIT's refractive surgery service for their preoperative examination. Eligibility for participation in the NG was confirmed by consecutive topographies, while all NG participants had to present uneventful ophthalmologic history, no indications of corneal pathology in slit-lamp biomicroscopy and Placido disk-based videokeratography.

INTERVENTIONS:
Procedure: Corneal Collagen Cross-linking (CXL) — Instillation of proparacaine hydrochloride 0.5% drops for topical anaesthesia, application of a sponge saturated with 10% alcohol to the central cornea for 20-30 seconds and subsequent de-epithelialization by means of a hockey knife. Following de-epithelialization, a mixture of 0.1% riboflavin in 20% Dextran solution was instilled to the cornea for 30 minutes (2 drops every 2 minutes) prior to the irradiation. In details, an 8.0mm diameter of central cornea was irradiated for 30 minutes by UVA light with a wavelength of 370nm and an irradiance of 3mW/cm2.The UVA radiation source that was used is the UV-XTM (IROC AG, Zurich, Switzerland). Instillation of riboflavin drops (1 drop every 2 minutes) was continued during irradiation, as well.
  Groups: Collagen-Cross-linking group (CXLG)

SUMMARY:
Primary objective of this study was to assess the intrasession, intersession and interobserver variability of the Pentacam-derived curvature and zernike coefficients in back surface of normal, keratoconic and crosslinked corneas.

DETAILED DESCRIPTION:
The Pentacam Classic (Oculus Optikgerate GmbH, Heidelberg, Germany, software version 1.14r04) was used for the sake of the study.Three study groups were formed: 1) Normal 2) Keratoconus group (KC) included patients with progressive keratoconus and 3) Collagen-Cross-linking group (CXL) included keratoconus patients that had been treated with uneventful CXL at least on year prior to their enrollment in the study.

Three consecutive scans were obtained by two experienced operators. The same procedure was repeated within two weeks for the assessment of intersession variability. In all cases acceptable maps had at least 10.0mm of corneal coverage. Keratometry (K), asphericity (Q), best-fit toric ellipsoid radius (Rs), eccentricity (ecc) and aberrometry (6.0mm pupil diameter), were analyzed. Furthermore we calculated and studied CRMS and CLRMS in order to better appreciate the visual significance of HOAs. Precision (Pre), repeatability (COR) and intraclass correlation coefficient (ICC), were calculated for evaluating intrasession and intersession repeatability. Bland-Altman analysis was used for assessing interobserver repeatability.

ELIGIBILITY:
Inclusion Criteria:

* Ideal refractive surgery candidate (Normal Group)
* Progressive keratoconus (Keratoconus group)
* Corneal collagen cross linking (CxL) treatment at least one year prior to enrollment (CxL group)

Exclusion Criteria:

(Normal Group)

* No indications of corneal pathology in slit-lamp biomicroscopy and Placido disk-based videokeratography
* Uneventful ophthalmologic history

All groups:

* Glaucoma
* Suspicion of glaucoma
* history of herpetic keratitis
* corneal scarring
* severe eye dryness
* pregnancy or nursing
* current corneal infection
* underlying autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from the Cornea service of the EIT in a consecutive-if-eligible basis.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Variability of posterior corneal surface curvature and aberrometric measurements within and between sessions and within and between observers. | 2 weeks
  The Pentacam Classic (Oculus Optikgerate GmbH, Heidelberg, Germany, software version 1.14r04) was used for the sake of the study. Three consecutive scans were obtained by two experienced operators for the assessment of intrasession and interobserver variability. The same procedure was repeated within two weeks for the assessment of intersession variability.Bland-Altman plots were used to evaluate agreement between the 2 operators. The reliability of all measurements was evaluated by means of the intraclass correlation coefficient(ICC).

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, Lecturer, Principal Investigator — Democritus University of Thrace
Locations (1):
- Eye Institute of Thrace (EIT), Alexandroupoli, Thrace, Greece